CLINICAL TRIAL: NCT00289965
Title: Brief Alcohol Interventions by Counselor vs Computer
Brief Title: Substance Use Risk Education (SURE) Project
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Kate B. Carey, PhD, Syracuse University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NIAAACAR012518-06; R01AA012518 (NIH); NIH Grant 2R01AA012518-06
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Alcohol Abuse; Alcohol Drinking
Keywords: Alcohol Abuse; Alcohol Drinking; Intervention Studies; Computer-Assisted Instruction; College Students
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): in-person brief motivational intervention
  Interventions: Behavioral: Counselor-administered Brief Motivational Intervention (BMI)
- 2 (Active Comparator): Alcohol 101plus
  Interventions: Behavioral: Alcohol 101 Plus (interactive CD-ROM)
- 3 (Active Comparator): AlcoholEdu (a Web-based tutorial).
  Interventions: Behavioral: AlcoholEdu (Internet-based tutorial)

INTERVENTIONS:
Behavioral: Counselor-administered Brief Motivational Intervention (BMI) — Students participate in a randomized study to evaluate 3 brief interventions: in-person brief motivational intervention, Alcohol 101plus (an interactive CD-ROM program), and AlcoholEdu (a Web-based tutorial). Participants will be followed over 12 months to determine changes in alcohol consumption and related problems.
  Arms: 1
Behavioral: Alcohol 101 Plus (interactive CD-ROM) — Students participate in a randomized study to evaluate 3 brief interventions: in-person brief motivational intervention, Alcohol 101plus (an interactive CD-ROM program), and AlcoholEdu (a Web-based tutorial). Participants will be followed over 12 months to determine changes in alcohol consumption and related problems.
  Arms: 2
Behavioral: AlcoholEdu (Internet-based tutorial) — Students participate in a randomized study to evaluate 3 brief interventions: in-person brief motivational intervention, Alcohol 101plus (an interactive CD-ROM program), and AlcoholEdu (a Web-based tutorial). Participants will be followed over 12 months to determine changes in alcohol consumption and related problems.
  Arms: 3

SUMMARY:
This project is designed to compare college drinking interventions on outcomes and cost-effectiveness. We plan to recruit 700 students with residence hall alcohol violations to participate in a randomized study to evaluate 3 brief interventions: in-person brief motivational intervention, Alcohol 101plus (an interactive CD-ROM program), and AlcoholEdu (a Web-based tutorial). Participants will be followed over 12 months to determine changes in alcohol consumption and related problems. We will also explore which participants might respond better to one intervention vs the others.

DETAILED DESCRIPTION:
Many college students engage in heavy episodic drinking, a pattern that increases risks of undesired academic, social, health, and legal consequences. Fortunately, brief motivational interventions - when administered during face-to-face sessions by a trained counselor - can help students to reduce their heavy drinking and related consequences. However, use of such counselor-administered interventions on college campuses remains infrequent; instead, administrators rely on computerized brief interventions because they can be administered with fewer staff at lower cost. Two computer-administered interventions (AlcoholEdu and Alcohol 101 Plus) are used by more than 1,000 colleges and universities nationwide, even though these interventions have not been evaluated in controlled studies. Despite the magnitude of the college-drinking problem, no data have addressed the differential efficacy (or cost-effectiveness) of the computer-administered versus counselor-administered brief motivational interventions. Thus, the primary purpose of the proposed research is to address gaps in the scientific literature by evaluating outcomes of three types of brief motivational interventions: a theoretically-based and empirically-tested counselor-administered intervention and the two most popular computerized interventions. A secondary purpose of the proposed research is to identify predictors of outcomes, and moderators associated with differential intervention response. A tertiary purpose is to assess the cost-effectiveness of three types of brief motivational interventions. The proposed research will be a randomized controlled trial with four treatment conditions and four assessment occasions. We will recruit at-risk student drinkers who have been sanctioned to receive an alcohol education intervention because they violated a residence hall policy. These referred students will be randomized to one of the three interventions, or to a delayed intervention control; and assessed at baseline and again 1, 6, and 12 months later on key drinking and drinking consequences outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Freshman, sophomore, and junior college students
* Students sanctioned for an alcohol-related violation on campus

Exclusion Criteria:

* Year in college: senior

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 703 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
mean number of drinks per week | 12 months
drinks per drinking day | 12 months
frequency of heavy drinking episodes | 12 months
peak blood alcohol concentration (BAC) | 12 months
Rutgers Alcohol Problems Index (RAPI) score | 12 months

SECONDARY OUTCOMES:
readiness to change | 12 months
decisional balance | 12 months
client satisfaction | 12 months
norms perception | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate B. Carey, PhD, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University, Syracuse, New York, United States

REFERENCES:
- [Derived] Fernandez AC, Yurasek AM, Merrill JE, Miller MB, Zamboanga BL, Carey KB, Borsari B. Do brief motivational interventions reduce drinking game frequency in mandated students? An analysis of data from two randomized controlled trials. Psychol Addict Behav. 2017 Feb;31(1):36-45. doi: 10.1037/adb0000239. Epub 2016 Dec 12. PMID 27936818
- See also: College Drinking: Changing the Culture - includes research, statistics, approaches to prevention, and interactive tools for students and educators. — http://www.collegedrinkingprevention.gov/